CLINICAL TRIAL: NCT01678313
Title: COX-2 Inhibitor Reduces Serum PSA Levels Might Predict a Lower Risk of Prostatic Cancer in Men With LUTS/BPH With an Elevated PSA Level
Brief Title: Cyclooxygenase-2 (COX-2) Inhibitor Reduces Serum Prostatic Specific Antigen (PSA) Levels
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Hann-Chorng Kuo, Department of Urology, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCGHUROL004
Record Dates: First submitted 2012-08-29; First posted 2012-09-05 (Estimated); Results first posted 2014-06-30 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign prostatic hyperplasia (BPH); Lower urinary tract symptoms (LUTS); Prostatic specific antigen (PSA); Cyclooxygenase-2 (COX-2)
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — Doxazosin; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study group (Experimental): Doxazosin 4 mg daily plus celecoxib 200 mg every day (QD)
  Interventions: Drug: Doxazosin 4 mg daily plus Celecoxib 200 mg every day (QD)
- Control group (Experimental): Doxazosin 4 mg every day (QD)
  Interventions: Drug: Doxazosin 4 mg every day (QD)

INTERVENTIONS:
Drug: Doxazosin 4 mg daily plus Celecoxib 200 mg every day (QD) — Study group
  Other Names: Doxazosin 4 mg; Celecoxib 200 mg
  Arms: Study group
Drug: Doxazosin 4 mg every day (QD) — Control group
  Other Names: Doxazosin 4 mg
  Arms: Control group

SUMMARY:
To investigate the therapeutic effect and safety of celecoxib adding on doxazosin and the potential predictive value of the absence of prostate cancer in the treatment of patients with LUTS/BPH and an elevated serum PSA level.

Patients who meet all eligible requirements for entry into the study will be randomized into one of the two treatment groups for 3 months in 2:1 ratio as shown below:

1. Doxazosin 4 mg daily plus celecoxib 200 mg every day (QD)
2. Doxazosin 4mg every day (QD)

DETAILED DESCRIPTION:
Study Procedure

* Male patients aged 40 years or older, having LUTS for at least 3 months (IPSS ≥ 8), a serum PSA level ≥ 4 ng/mL, without a palpable prostatic nodule will be enrolled into this prospective randomized trial to investigate whether COX-2 inhibitor can decrease serum PSA level and acts as a biomarker to differentiate between chronic inflammation and prostate cancer.
* Eligible subjects will be randomly assigned to the study and control groups at 2:1 ratio. The study group will receive doxazosin 4mg every day (QD) plus celecoxib 200mg QD for 3 months and the control group will receive doxazosin 4 mg QD for 3 months. Patients will be investigated for IPSS, total prostatic volume, transition zone index, maximum flow rate, voided volume, postvoid residual, serum PSA, free PSA and serum C-reactive protein (CRP) levels at baseline and 3 months after treatment. If the serum PSA levels remained higher than 4 ng/mL, patients of either group will be advised to receive prostatic biopsy for histopathological investigation.
* The prostatic biopsy will be advised at the end of the study in both groups of patients. Ten prostatic biopsied strips will be sent to pathological department for investigating the existence of prostatic cancer. The other two strips will be stored in liquid nitrogen for further investigation of inflammatory biomarkers.

Data Analysis

* The efficacy evaluation will be performed on intention-to-treat populations (ITT) and per-protocol populations (PPP) datasets while the safety evaluation will be performed on ITT datasets. The primary conclusion will be made for the primary endpoint and secondary endpoint on the ITT population.

Efficacy Endpoint Analysis

* Net change of each efficacy item will be analyzed by paired t-test between baseline and post-treatment in the treatment group and controlled group. The net changes of each efficacy item will be analyzed by ANOVA test to compare between treatment group and controlled group. The global assessment by the patients will be analyzed by chi-square test between the treatment and controlled group.
* All efficacy variables will be reported of respective point estimated and 95% confidence interval. Comparison tests will be reported of respective p value.

Safety Endpoints

* Adverse events will be reported by both controlled and treatment groups and by physiological systems as appropriate. Incidence of adverse events and the categories of adverse event severity between treatments will be analyzed by Cochran-Mantel-Haenszel test. The coding system used will be the Coding Symbols for a Thesaurus of Adverse Reaction Terms (COSTART).

Changes in physical examinations will be displayed for each individual system.

* All statistical tests used will be two-tailed with α= 0.05.

Expected Results and Conclusion

* Chronic inflammation has been considered a possible but important factor to induce LUTS and promote prostatic growth. PSA elevation is a sensitive but not specific sign for prostatic cancer. In order to reduce the need for prostatic biopsy in patients with an elevated serum PSA level, the results of this study might provide a simple way for initial differential diagnosis of chronic inflammation from prostatic cancer. If serum PSA can be reduced significantly after celecoxib therapy and the positive biopsy rate of the following prostatic biopsy is lower than the control group, we might use this treatment for the initial management of high PSA level in men with LUTS/BPH. Furthermore, if chronic inflammation of the prostate can be reduced, the bothersome of the LUTS as well as voiding condition might be improved. This result can be another benefit for men who are suffering from LUTS and worried about surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male adults aged ≥ 40 years with LUTS/BPH, IPSS ≥ 8
* Free of active urinary tract infection
* Free of neurogenic voiding dysfunction
* No history of previous prostate biopsy within 6 months
* No treatment of BPH by alpha-blocker or 5-alpha-reductase inhibitor within 6 months
* Patient or his legally acceptable representative has signed the written informed consent form

Exclusion Criteria:

* Patients with severe cardiopulmonary disease and such as congestive heart failure, arrhythmia, poorly controlled hypertension, not able to receive regular follow-up
* Patients with acute r chronic urinary retention and urodynamically proven detrusor underactivity
* Patients with postvoid residual > 250 mL
* Patients have laboratory abnormalities at screening including:

  1. Aspartate aminotransferase (AST) > 3 x upper limit of normal range
  2. Alanine aminotransferase (ALT) > 3 x upper limit of normal range
  3. Patients have abnormal serum creatinine level > 2 x upper limit of normal range
* Patients with any other serious disease or condition considered by the investigator not suitable for entry into the trial
* Patients participated investigational drug trial within 1 month before entering this study

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hann-Chorng Kuo, M.D., Principal Investigator — Department of Urology, Buddhist Tzu Chi General Hospital and Tzu Chi University
Locations (1):
- Buddhist Tzu Chi General Hospital, Hualien City, Taiwan

REFERENCES:
- [Background] Liu HT, Kuo HC. Urinary nerve growth factor levels are increased in patients with bladder outlet obstruction with overactive bladder symptoms and reduced after successful medical treatment. Urology. 2008 Jul;72(1):104-8; discussion 108. doi: 10.1016/j.urology.2008.01.069. Epub 2008 Apr 8. PMID 18400272
- [Background] St Sauver JL, Sarma AV, Jacobson DJ, McGree ME, Lieber MM, Girman CJ, Nehra A, Jacobsen SJ. Associations between C-reactive protein and benign prostatic hyperplasia/lower urinary tract symptom outcomes in a population-based cohort. Am J Epidemiol. 2009 Jun 1;169(11):1281-90. doi: 10.1093/aje/kwp085. Epub 2009 Apr 24. PMID 19395697
- [Background] Andersson KE. LUTS treatment: future treatment options. Neurourol Urodyn. 2007 Oct;26(6 Suppl):934-47. doi: 10.1002/nau.20500. PMID 17696154
- [Background] Kuo HC. Videourodynamic analysis of pathophysiology of men with both storage and voiding lower urinary tract symptoms. Urology. 2007 Aug;70(2):272-6. doi: 10.1016/j.urology.2007.03.063. PMID 17826488
- [Background] Di Silverio F, Gentile V, De Matteis A, Mariotti G, Giuseppe V, Luigi PA, Sciarra A. Distribution of inflammation, pre-malignant lesions, incidental carcinoma in histologically confirmed benign prostatic hyperplasia: a retrospective analysis. Eur Urol. 2003 Feb;43(2):164-75. doi: 10.1016/s0302-2838(02)00548-1. PMID 12565775
- [Background] Sciarra A, Mariotti G, Salciccia S, Autran Gomez A, Monti S, Toscano V, Di Silverio F. Prostate growth and inflammation. J Steroid Biochem Mol Biol. 2008 Feb;108(3-5):254-60. doi: 10.1016/j.jsbmb.2007.09.013. Epub 2007 Sep 7. PMID 17935971
- [Background] Sciarra A, Di Silverio F, Salciccia S, Autran Gomez AM, Gentilucci A, Gentile V. Inflammation and chronic prostatic diseases: evidence for a link? Eur Urol. 2007 Oct;52(4):964-72. doi: 10.1016/j.eururo.2007.06.038. Epub 2007 Jul 2. PMID 17618043
- [Background] Alcaraz A, Hammerer P, Tubaro A, Schroder FH, Castro R. Is there evidence of a relationship between benign prostatic hyperplasia and prostate cancer? Findings of a literature review. Eur Urol. 2009 Apr;55(4):864-73. doi: 10.1016/j.eururo.2008.11.011. Epub 2008 Nov 21. PMID 19027219
- [Background] Di Silverio F, Bosman C, Salvatori M, Albanesi L, Proietti Pannunzi L, Ciccariello M, Cardi A, Salvatori G, Sciarra A. Combination therapy with rofecoxib and finasteride in the treatment of men with lower urinary tract symptoms (LUTS) and benign prostatic hyperplasia (BPH). Eur Urol. 2005 Jan;47(1):72-8; discussion 78-9. doi: 10.1016/j.eururo.2004.08.024. PMID 15582252
- [Background] Ozdemir I, Bozkurt O, Demir O, Aslan G, Esen AA. Combination therapy with doxazosin and tenoxicam for the management of lower urinary tract symptoms. Urology. 2009 Aug;74(2):431-5. doi: 10.1016/j.urology.2009.01.088. Epub 2009 Jun 7. PMID 19501883
- [Background] Jang J, Park EY, Seo SI, Hwang TK, Kim JC. Effects of intravesical instillation of cyclooxygenase-2 inhibitor on the expression of inducible nitric oxide synthase and nerve growth factor in cyclophosphamide-induced overactive bladder. BJU Int. 2006 Aug;98(2):435-9. doi: 10.1111/j.1464-410X.2006.06207.x. PMID 16879691
- [Background] Falahatkar S, Mokhtari G, Pourreza F, Asgari SA, Kamran AN. Celecoxib for treatment of nocturia caused by benign prostatic hyperplasia: a prospective, randomized, double-blind, placebo-controlled study. Urology. 2008 Oct;72(4):813-6. doi: 10.1016/j.urology.2008.04.069. Epub 2008 Aug 9. PMID 18692876
- [Background] Djavan B, Waldert M, Zlotta A, Dobronski P, Seitz C, Remzi M, Borkowski A, Schulman C, Marberger M. Safety and morbidity of first and repeat transrectal ultrasound guided prostate needle biopsies: results of a prospective European prostate cancer detection study. J Urol. 2001 Sep;166(3):856-60. PMID 11490233

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 140 Patients with lower urinary tract symptoms (LUTS)/benign prostatic hyperplasia (BPH) and PSA>4 ng/dL underwent randomization 70 patients in study group 70 patients in control group
Period: Completed the 3-month Therapy
Arm/Group | Study Group | Control Group
Started | 70 | 70
Completed | 64 | 58
Not Completed | 6 | 12
Not completed — Lost to Follow-up | 3 | 8
Not completed — Physician Decision | 3 | 4
Period: PSA >4 ng/dL at 3 Months
Arm/Group | Study Group | Control Group
Started | 64 | 58
Completed | 56 | 49
Not Completed | 8 | 9
Not completed — PSA≦4 | 8 | 9
Period: Prostate Biopsy at 3 Months
Arm/Group | Study Group | Control Group
Started | 56 | 49
Completed | 45 | 37
Not Completed | 11 | 12
Not completed — Not received prostate biopsy | 11 | 12

BASELINE CHARACTERISTICS:
Groups:
- Study Group: Doxazosin 4 mg daily plus celecoxib 200 mg daily, complete 3 month therapy N=64(91.4%)
- Control Group: Doxazosin 4 mg alone everyday, complete 3 month therapy N=58(82.9%)
- Total: Total of all reporting groups
Arm/Group | Study Group | Control Group | Total
Number analyzed (Participants) | 64 | 58 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.4 (9.5) | 73.8 (8.0) | 72.1 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 64 | 58 | 122
Region of Enrollment [Number; unit: participants]
  Taiwan | 64 | 58 | 122

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Serum Prostate Specific Antigen (PSA) Level
Description: Efficacy:
  Change from Baseline in the serum PSA level from baseline and 3 months Change = Month 3 minus Baseline value
Time Frame: Baseline and 3 months after initial treatment
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 45 | 37
ng/mL
  Baseline | 10.8 (5.42) | 15.2 (12.7)
  3 months | 9.42 (5.41) | 13.5 (10.6)
  Change | -1.43 (0.01) | -1.70 (2.15)

2. Secondary Outcome: Change From Baseline in the Void Volume (VV)
Description: Efficacy:
  Change from Baseline in the Void Volume (VV) from baseline and 3 months Change = Month 3 minus Baseline value
Time Frame: Baseline and 3 months after initial treatment
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 45 | 37
mL
  Baseline | 259 (113) | 175 (107)
  3 months | 227 (80.8) | 231 (134)
  Change | -32.3 (32.1) | 55.7 (27.3)

3. Secondary Outcome: Change From Baseline in the Maximum Flow Rate (Qmax)
Description: Efficacy:
  Change from Baseline in the maximum flow rate (Qmax) from baseline and 3 months Change = Month 3 minus Baseline value
Time Frame: Baseline and 3 months after initial treatment
Measure: Mean (Standard Deviation); unit: mL/s
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 45 | 37
mL/s
  Baseline | 12.2 (4.67) | 10.0 (6.2)
  3 months | 12.2 (4.19) | 11.9 (6.61)
  Change | -0.09 (0.49) | 1.9 (0.41)

4. Secondary Outcome: Change From Baseline in the IPSS Subscore (IPSS Voiding) Questionnaires
Description: Efficacy:
  Change from Baseline in the IPSS Voiding from baseline and 3 months. The IPSS subscore (IPSS Voiding) questionnaires is a 4 symptom questions. The symptom score have 6-point scale ranging from 0 "Not at all" to 5 "Almost always". Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom.
  The total IPSS Voiding score can therefore range from 0 to 20 (asymptomatic to very symptomatic).
  Change = Month 3 minus Baseline value
Time Frame: Baseline and 3 months after initial treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 45 | 37
units on a scale
  Baseline | 7.55 (6.84) | 5.54 (5.12)
  3 months | 3.84 (4.57) | 3.45 (4.22)
  Change | -3.71 (2.27) | -2.09 (0.9)

5. Secondary Outcome: Change From Baseline in the IPSS Subscore (IPSS Storage) Questionnaires
Description: Efficacy:
  Change from Baseline in the IPSS Storage from baseline and 3 months The IPSS subscore (IPSS Storage) is a 3 symptom questions. The symptom score have 6-point scale ranging from 0 "Not at all" to 5 "Almost always". Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom.
  The total IPSS Storage score can therefore range from 0 to 15 (asymptomatic to very symptomatic).
  Change = Month 3 minus Baseline value
Time Frame: Baseline and 3 months after initial treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 45 | 37
units on a scale
  Baseline | 5.59 (3.72) | 6.06 (3.38)
  3 months | 3.09 (1.4) | 4.01 (2.04)
  Change | -2.5 (2.32) | -2.05 (1.34)

6. Secondary Outcome: Change From Baseline in the International Prostate Symptom Score (IPSS) Questionnaires
Description: Efficacy:
  Change from Baseline in the International Prostate Symptom Score (IPSS) from baseline and 3 months The International Prostate Symptom Score (IPSS) is an 7 symptom questions including 4 voiding questions (IPSS Voiding), 3 storage questions (IPSS Storage) The symptom score have 6-point scale ranging from 0 "Not at all" to 5 "Almost always".
  Total IPSS score = IPSS voiding + IPSS Storage Rang = 0 to 35 (asymptomatic to very symptomatic). Mild = 0 to 7; Moderate = 8 to 19; Severe = 20 to 35
  Change = Month 3 minus Baseline value
Time Frame: Baseline and 3 months after initial treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 45 | 37
units on a scale
  Baseline | 13.1 (7.65) | 12.0 (7.65)
  3 months | 6.45 (3.18) | 7.70 (5.11)
  Change | -6.63 (4.47) | -4.31 (2.54)

ADVERSE EVENTS:
Time Frame: During the 3-month clinical follow up
Description: No patient suffered from heart attack, stroke, thromboembolic events or peptic ulcer. No adverse event related to the test medications was observed.
Arm/Group | Study Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/58
Other Adverse Events (participants affected / at risk) | 0/64 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes